CLINICAL TRIAL: NCT03976128
Title: Effect of Nordic Walking Training Compared With Conventional Endurance Training in Walking Capacity in People With Multiple Sclerosis: a Simple Blinded Randomized Controlled Trial
Brief Title: Endurance and Walking Training by Nordic Walking in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Multiple Sclerosis Center of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nordic Walking in MS
Record Dates: First submitted 2019-06-01; First posted 2019-06-05 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
Keywords: endurance training; nordic walking; walking ability; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic Walking training (Experimental): 20 sessions of 45 minutes x 2 times/week x 10 weeks using NW
  Interventions: Behavioral: Nordic Walking Training
- Conventional endurance training (Active Comparator): 20 sessions of 45 minutes x 2 times/week x 10 weeks using treadmill and cycloergometer training.
  Interventions: Behavioral: Conventional endurance training

INTERVENTIONS:
Behavioral: Nordic Walking Training — The excursions will take place predominantly in flat pathways, beginning in a local park and progressing to roadside footpaths. Each session will last an hour including a warm up, NW and a cool down with stretching exercises.
  Arms: Nordic Walking training
Behavioral: Conventional endurance training — 15 minutes of Treadmill training with progressive increase of velocity followed by 20 minutes of cycloergometer with progressive increase of resistance. Each session will last an hour including a warm up, training with treadmill and cycloergometer and a cool down with stretching exercises.
  Arms: Conventional endurance training

SUMMARY:
Walking capacity is one of the most valuable body functions among persons with multiple sclerosis (MS) and it is one of the most frequently affected, even in early stages of the disease. Inactivity and deconditioning can accelerate gait impairment and promote other pathologies related with sedentary lifestyle.

Nordic walking (NW) is a fun and effective fitness and rehabilitation activity. The benefits of NW have been extensively described in healthy and elderly population (Tschentscher, 2013; Kappor, 2013) and it is proving to be highly recommended to different neurological conditions, specially to Parkinson Disease (Reuter 2006; van Eijkeren 2008; Fritz 2011; Ebersbach 2014).

There is no evidence on NW and MS, although it's supposed to be an ideal physical activity for many reasons: it tones the upper and lower body at the same time, uses 90% of the skeletal muscles, burns up to 46% more calories than ordinary walking, reduces the pressure on knees and joints, poles propel the walker along easier and faster and it is one of the most effective cross training techniques for people who require improve cardiovascular and endurance conditioning.

DETAILED DESCRIPTION:
A simple blinded randomized controlled trial as designed to assess if an endurance training (20 sessions of 45 minutes x 2 times/week x 10 weeks) using NW improves: walking capacity, balance, fatigue, mood and health-related quality of life of people with MS.

66 people with MS will be randomly allocated in NW group or conventional endurance training group (treadmill and cycloergometer). Assessments will take place before starting the training, after the training and 3 months after.

ELIGIBILITY:
Inclusion Criteria:

* People over 18 diagnosed of MS following the Mc Donald criteria, clinically stable who:
* show mild to moderate balance disorder (BBS>45). Mild risk of falls.
* refer fatigue during walking and restriction on their usual walking distance during the last 6 months.
* Accept to participate in the study and signed the informed consent.

Exclusion Criteria:

* Other neurological disorders.
* Moderate to severe spasticity (Ashworth>2)
* Non stable heart diseases, diabetes mellitus, arthritis in lower limbs, acute pain in lower limbs, peripheral neuropathies, severe orthopedics problems, psychiatric problems, pregnancy.
* Incapacity to maintain a minimum walking rhythm at least during 15 minutes.
* Cognitive disability or body schema disorder that limits to fill in the assessment questionaires or understanding and applying the technique.
* To be training in other physical activities that can modify the level of fatigue or walking ability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test (6MWT) | Assessment will take place at baseline and after 10 weeks
  Maximal distance (in meters) walked during 6 minutes
Change from baseline 6 Minute Walk Test (6MWT) to 6 months | Assessment will take place up to 6 months, through the study completion
  Maximal distance (in meters) walked during 6 minutes

SECONDARY OUTCOMES:
Timed 25 Foot Walk Test | Assessment will take place at baseline and after 10 weeks
  The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
Change from baseline Timed 25 Foot Walk Test to 6 months | Assessment will take place up to 6 months, through the study completion
  The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.
Multiple Sclerosis Walking Scale 12 | Assessment will take place at baseline and after 10 weeks
  12-item self reported measure of the impact of MS on individual's walking ability. Each item scoring provides options 1-5, with 1 meaning no limitation and 5 meaning extreme limitation on the gait related item. The total score ranges between 12 and 60, with higher scores indicating more limitation perceived on walking ability.
Change from baseline Multiple Sclerosis Walking Scale 12 to 6 months | Assessment will take place up to 6 months, through the study completion
  12-item self reported measure of the impact of MS on individual's walking ability. Each item scoring provides options 1-5, with 1 meaning no limitation and 5 meaning extreme limitation on the gait related item. The total score ranges between 12 and 60, with higher scores indicating more limitation perceived on walking ability.
Timed Up and Go Test | Assessment will take place at baseline and after 10 weeks
  Time in seconds required to walk to a line that is 3 meters (9.8 feet) away, turn around at the line, walk back to the chair, and sit down.
Change from baseline Timed Up and Go Test to 6 months | Assessment will take place up to 6 months, through the study completion
  Time in seconds required to walk to a line that is 3 meters (9.8 feet) away, turn around at the line, walk back to the chair, and sit down.
Berg Balance Scale | Assessment will take place at baseline and after 10 weeks
  The Berg Balance Scale (BBS)14-item objective measure that assesses static balance and fall risk in adults. Items include static and dynamic activities with varying difficulty. Each item scoring provides options 0-4, determined by the ability to perform the assessed ability. Item score are then summed ranging between 12 and 60, with higher scores indicating better balance ability
Change from baseline Berg Balance Scale to 6 months | Assessment will take place up to 6 months, through the study completion
  The Berg Balance Scale (BBS)14-item objective measure that assesses static balance and fall risk in adults. Items include static and dynamic activities with varying difficulty. Each item scoring provides options 0-4, determined by the ability to perform the assessed ability. Item score are then summed ranging between 12 and 60, with higher scores indicating better balance ability
Activities Specific Balance Confidence Scale | Assessment will take place at baseline and after 10 weeks
  The Activities Specific Balance Confidence Scale(ABC scale) is a reported measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. The scale has 16 items (score 0-1600 possible). The score is recorded as a percentage (%), with 100% the highest level of confidence. Max score of 1600 divided by 16 items = 100%
Change from baseline Activities Specific Balance Confidence Scale to 6 months | Assessment will take place up to 6 months, through the study completion
  The Activities Specific Balance Confidence Scale(ABC scale) is a reported measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. The scale has 16 items (score 0-1600 possible). The score is recorded as a percentage (%), with 100% the highest level of confidence. Max score of 1600 divided by 16 items = 100%
Modified Fatigue Impact Scale | Assessment will take place at baseline and after 10 weeks
  The Modified Fatigue Impact Scale (MFIS) is a form of the Fatigue Impact Scale (Fisk et al, 1994) based on items derived from interviews with MS patients concerning how fatigue interferes in their lifes. The instrument provides an assessment of the effect of fatigue in terms of physical, mental and psychosocial functioning. Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities. The Physical Subscale range from 0 to 36. The Cognitive Subscale ranges from 0 to 40. The Psychosocial Subscale ranges from 0 to 8.The total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales.
Change from baseline Modified Fatigue Impact Scale to 6 months | Assessment will take place up to 6 months, through the study completion
  The Modified Fatigue Impact Scale (MFIS) is a form of the Fatigue Impact Scale (Fisk et al, 1994) based on items derived from interviews with MS patients concerning how fatigue interferes in their lifes. The instrument provides an assessment of the effect of fatigue in terms of physical, mental and psychosocial functioning. Items on the MFIS can be aggregated into three subscales (physical, cognitive, and psychosocial), as well as into a total MFIS score. All items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities. The Physical Subscale range from 0 to 36. The Cognitive Subscale ranges from 0 to 40. The Psychosocial Subscale ranges from 0 to 8.The total MFIS score can range from 0 to 84. It is computed by adding scores on the physical, cognitive, and psychosocial subscales.
Multiple Sclerosis Quality of Life 54 | Assessment will take place at baseline and after 10 weeks
  The Multiple Sclerosis Quality of Life 54 (MSQoL-54) is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The summary scores are the physical health composite summary and the mental health composite summary, that are derived from a weighted combination of scale scores. Higher scores means better quality of life perceived.
Change from baseline Multiple Sclerosis Quality of Life 54 to 6 months | Assessment will take place up to 6 months, through the study completion
  The Multiple Sclerosis Quality of Life 54 (MSQoL-54) is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. This 54-item instrument generates 12 subscales along with two summary scores, and two additional single-item measures. The subscales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The summary scores are the physical health composite summary and the mental health composite summary, that are derived from a weighted combination of scale scores. Higher scores means better quality of life perceived.

CONTACTS AND LOCATIONS:
Overall Officials: Carme Santoyo Medina, PT, MSc, Principal Investigator — Multiple Sclerosis Center of Catalonia
Locations (1):
- Multiple Sclerosis Center of Catalonia, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vidal-Jordana A, Montalban X. Multiple Sclerosis: Epidemiologic, Clinical, and Therapeutic Aspects. Neuroimaging Clin N Am. 2017 May;27(2):195-204. doi: 10.1016/j.nic.2016.12.001. PMID 28391781
- [Background] de Sa J. [Epidemiology of multiple sclerosis in Portugal and Spain]. Rev Neurol. 2010 Oct 1;51(7):387-92. No abstract available. Spanish. PMID 20859919
- [Background] Otero S, Batlle J, Bonaventura I, Brieva L, Bufill E, Cano A, Carmona O, Escartin A, Marco M, Moral E, Munteis E, Nos C, Pericot I, Perkal H, Ramio-Torrenta L, Ramo-Tello C, Saiz A, Sastre-Garriga J, Tintore M, Vaque J, Montalban X; Grupo de Trabajo del Registro de Esclerosis Multiple de Cataluna. [Multiple sclerosis epidemiological situation update: pertinence and set-up of a population based registry of new cases in Catalonia]. Rev Neurol. 2010 May 16;50(10):623-33. Spanish. PMID 20473839
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Tallner A, Waschbisch A, Wenny I, Schwab S, Hentschke C, Pfeifer K, Maurer M. Multiple sclerosis relapses are not associated with exercise. Mult Scler. 2012 Feb;18(2):232-5. doi: 10.1177/1352458511415143. Epub 2011 Jul 6. PMID 21733890
- [Result] Motl RW, McAuley E, Snook EM. Physical activity and multiple sclerosis: a meta-analysis. Mult Scler. 2005 Aug;11(4):459-63. doi: 10.1191/1352458505ms1188oa. PMID 16042230
- [Result] Rietberg MB, Brooks D, Uitdehaag BM, Kwakkel G. Exercise therapy for multiple sclerosis. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003980. doi: 10.1002/14651858.CD003980.pub2. PMID 15674920
- [Result] Motl RW, Fernhall B, McAuley E, Cutter G. Physical activity and self-reported cardiovascular comorbidities in persons with multiple sclerosis: evidence from a cross-sectional analysis. Neuroepidemiology. 2011;36(3):183-91. doi: 10.1159/000327749. Epub 2011 May 20. PMID 21597305
- [Result] Dalgas U, Stenager E, Ingemann-Hansen T. Multiple sclerosis and physical exercise: recommendations for the application of resistance-, endurance- and combined training. Mult Scler. 2008 Jan;14(1):35-53. doi: 10.1177/1352458507079445. Epub 2007 Sep 19. PMID 17881393
- [Result] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Fatigue, mood and quality of life improve in MS patients after progressive resistance training. Mult Scler. 2010 Apr;16(4):480-90. doi: 10.1177/1352458509360040. Epub 2010 Mar 1. PMID 20194584
- [Result] Newman MA, Dawes H, van den Berg M, Wade DT, Burridge J, Izadi H. Can aerobic treadmill training reduce the effort of walking and fatigue in people with multiple sclerosis: a pilot study. Mult Scler. 2007 Jan;13(1):113-9. doi: 10.1177/1352458506071169. PMID 17294619
- [Result] Mostert S, Kesselring J. Effects of a short-term exercise training program on aerobic fitness, fatigue, health perception and activity level of subjects with multiple sclerosis. Mult Scler. 2002 Apr;8(2):161-8. doi: 10.1191/1352458502ms779oa. PMID 11990874
- [Result] Weikert M, Dlugonski D, Balantrapu S, Motl RW. Most common types of physical activity self-selected by people with multiple sclerosis. Int J MS Care. 2011 Spring;13(1):16-20. doi: 10.7224/1537-2073-13.1.16. PMID 24453701
- [Result] McAuley E, Motl RW, Morris KS, Hu L, Doerksen SE, Elavsky S, Konopack JF. Enhancing physical activity adherence and well-being in multiple sclerosis: a randomised controlled trial. Mult Scler. 2007 Jun;13(5):652-9. doi: 10.1177/1352458506072188. Epub 2007 Feb 9. PMID 17548446
- [Result] Dettmers C, Sulzmann M, Ruchay-Plossl A, Gutler R, Vieten M. Endurance exercise improves walking distance in MS patients with fatigue. Acta Neurol Scand. 2009 Oct;120(4):251-7. doi: 10.1111/j.1600-0404.2008.01152.x. Epub 2009 Jan 28. PMID 19178385
- [Result] Pilutti LA, Platta ME, Motl RW, Latimer-Cheung AE. The safety of exercise training in multiple sclerosis: a systematic review. J Neurol Sci. 2014 Aug 15;343(1-2):3-7. doi: 10.1016/j.jns.2014.05.016. Epub 2014 May 15. PMID 24880538